CLINICAL TRIAL: NCT05309031
Title: An Immersion Intervention for Symptoms of PTSD in Student Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Rebecca Benfield, Principal Investigator, University of Nevada, Las Vegas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNevada
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Single group repeated measures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immersion (Experimental): This group will receive the immersion intervention
  Interventions: Other: Water Immersion

INTERVENTIONS:
Other: Water Immersion — Participants will enter the pool, which has a thermoneutral temperature of 33°C (92°F), warm enough to be comfortable, but cool enough to avoid an increase in HR with similar ambient air temperature. A maximum depth of 4 to 4 feet 6 inches allows ample room participants to be immersed to the chest, float vertically and move in the pool. During 45 min of immersion, they will be instructed to stand, walk and move ad lib. Noodles will be available to hang or rest on in a vertical position. Taller participants will remain at the pool's deep end. The timeframe was chosen to approximate our previous immersion intervention length.

SUMMARY:
This study will explore the physical and psychological effects of warm water immersion to the chest on student Veterans who experience symptoms of Post-Traumatic Stress Disorder (PTSD) and may also have depression, anxiety and pain.

DETAILED DESCRIPTION:
Procedure/Protocol

Data collection will occur over 15+ consecutive weeks depending on recruitment success and scheduling availability of participants.

Day 1: After reviewing, answering questions and signing the consent form with the PI (5-20 min) , demographic information will be collected, the PCL-5 (10 min), PHQ-9 (10 min) and CES scale (5 min) will be administered by a clinical psychologist or psychiatric nurse practitioner in a private room at the SON Research Office using paper instruments.

Day 2: Data will be collected on one participant at each session at the same time of the day to control for circadian rhythms in salivary sAA, using Salimetrics protocols: 1. Collection Methods: SalivaBio Oral Swab and 2. Collecting Salivary Amylase (Appendix 11 Swab, Appendix 12 Collection). Data will be collected at the Centennial Hills YMCA and includes these activities:

Salivary Amylase

* Avoid foods with high sugar or acidity, immediately before sample collection, since they may compromise the assay by lowering saliva pH and increasing bacterial growth.
* Document consumption of alcohol, caffeine, nicotine, and prescription/over-the-counter medications within the prior 12 hours.
* Medications that specifically agonize or antagonize alpha- or beta-adrenergic processes should be avoided
* Document vigorous physical activity and the presence of oral diseases or injury.
* Consider documenting parameters to estimate saliva flow rate.
* Rinse mouth with water to remove food residue and wait at least 10 minutes after rinsing to avoid sample dilution before collecting saliva.

Protocol After arrival at the YMCA, participants will remain seated for 10 min in a quiet room adjacent to the pool area. Then pencil and paper instruments (VASA [20 sec], VASP [20 sec], MDMQ [ 7min]) will be administered and sAA collected (5min) by the PI . Next, participants will change into swimwear and enter the pool (Appendix 13 Pool Photo). A timer will be set for 15 and 45 min of immersion, with the same sequence of data collected while participants are in the water. A lifeguard will be in attendance. Following completion of the immersion intervention, participants will get dressed in the adjacent locker room and be escorted to a private room adjacent to the pool area where individual interviews will be conducted (30-60 min).

All participants are able to withdraw from the study at any time. If data has been collected on day 1 and on day 2 at baseline and 15 minutes it will be retained and analyzed.

An interview guide consisting of questions related to the intervention and participant cues will direct the conversation (Appendix 10 Interview Questions).

The interview will be initiated using a grand tour question, such as "Tell me about your experience while immersed in the water. How did you feel?" then proceed to more directed questions related to specific symptoms and specific emotional and psychological responses to the intervention (immersion). Participants may be asked to expand on specific items as applicable. At the conclusion, the participant will be asked if they have any questions or if there is anything else they would like to add. All interviews will be audio-recorded and transcribed, however, if any participants do not consent to be recorded, the researcher will take notes. Participants may conclude the interview at any time, and should they experience distress or strong emotions, the interview will be terminated. All participants will be provided with a list of available support resources.

Semi-structured interview and audio recording of the interview will be conducted in a private conference room. Only participant code numbers will be included. The audio recording on the digital recorder will never leave the investigator's presence and will be saved to the investigator's desktop on a private, pass coded protected UNLV computer, housed in a locked room. The audio recording will be immediately saved to the secure UNLV google shared drive and immediately deleted from the digital recorder and the computer desktop.

Before beginning the interview, participants will be informed that the meeting is being recorded prior to beginning the conversation. They will also be informed that the audio recording of the interview is being saved for analysis. Participants will be informed that a "code number" will be used during the interview to protect their identity.

A certified transcriptionist service Rev.com will transcribe the digitally audio recorded interview data verbatim. Rev.com has an established transcriber confidentiality agreement signed by all transcriptionists. The digitally audio recorded interview will be labeled with unique anonymous code number identifier and securely digitally delivered to the transcribing service. Transcribed transcripts will not contain personal identifying information about the participant. Once the audio recording has been converted to text, the recording residing on the secure UNLV google shared drive will be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of previous military service, current enrollment as a student at UNLV, and current PTSD symptoms. They must be able to enter and exit the pool without assistance.

Exclusion Criteria:

* Self-report of current dental, cardiac, pulmonary or kidney disease, uncontrolled diabetes, HIV, hepatitis, mental illness (except depression), traumatic brain injury, morbid obesity, open wounds, fear of water, or missing lower extremities and presumptive or confirmed pregnancy. Pharmacologics, including antidepressants, analgesics and non-steroidal anti-inflammatories, will not be controlled for because of the difficulty of recruiting participants without comorbid depression or pain.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Salivary Alpha-Amylase change is being assessed | Pre Immersion Baseline (dry) Immersion at 15 minutes (wet) and 45 minutes (wet)
  Salivary alpha-amylase samples will be analyzed by Salametrics, Carlsbad, CA using a Saliva Bio Oral Swab device and Swab Storage Tube, immediately placed on ice and frozen within 2 hours at -70 degrees. Frozen sample aliquots containing at least 325µL, will be shipped at one time, on dry ice for analysis using .25 µL, by a Kinetic Reaction assay, with a sensitivity of 0.4 U/ml, range of 2 - 400 U/ml. Samples are run in duplicate.
Multidimensional Mood State Questionnaire (MDMQ) Change is being assessed | Pre Immersion Baseline (dry) Immersion at 15 minutes (wet) and 45 minutes (wet)
  The Multidimensional Mood State Questionnaire (MDMQ) is an English version of the German Multidimensional Mood State Questionnaire. It is based on the condition diagnosis of three mood dimensions "elevated-depressed" (German) "good-bad" (English), (G Scale) "wakefulness drowsiness" (German) "awake-tired" (W Scale) and "restlessness" (German) "calm-nervous" (R scale) and considers situational effects. The reliabilities at four measurement times using split-half correlation with subsequent Spearman-Brown test extension calculation of the German version are G scale between .96 and .97, W scale between .94 and .96 and R scale between .87 and .94 (Steyer et al., 1994). Dr. Rolf Steyer confirms the scale has not been tested in English (personal communication). This scale is simple, easy to use and measures current mood.
Visual Analogue Scale (VAS) for Anxiety Change is being assessed | Pre Immersion Baseline (dry) Immersion at 15 minutes (wet) and 45 minutes (wet)
  Visual Analogue Scale (VAS) will measure anxiety. VAS reliability, validity, administration and scoring for anxiety and pain have been previously described (Benfield et al., 2001).Scores range between 0 and 100 mm. Lower scores mean less anxiety.
Visual Analogue Scale (VAS) for Pain Change is being assessed | Pre Immersion Baseline (dry) Immersion at 15 minutes (wet) and 45 minutes (wet)
  Visual Analogue Scale (VAS) will measure pain. VAS reliability, validity, administration and scoring for anxiety and pain have been previously described (Benfield et al., 2001)Scores range between 0 and 100 mm. Lower scores mean less pain.
Semi-structured interview | Immediately following immersion
  Individual semi-structured interviews will be completed to explore participant's overall perceptions of the immersion intervention and its effect on their general well-being and symptoms. Interviews will be conducted in a conversational tone, using open-ended questions, and active listening techniques. An interview guide consisting of questions related to the intervention and participant cues will direct the conversation The interview will be initiated using a grand tour question, such as "Tell me about your experience while immersed in the water. How did you feel?" then proceed to more directed questions related to specific symptoms related to specific emotional and psychological responses to the intervention (immersion). All interviews will be audio-recorded and transcribed, however, if any participants do not consent to be recorded, the researcher will take notes. Interviews are expected to take approximately 30 - 60 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Benfield, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- UNLV, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benfield RD, Hortobagyi T, Tanner CJ, Swanson M, Heitkemper MM, Newton ER. The effects of hydrotherapy on anxiety, pain, neuroendocrine responses, and contraction dynamics during labor. Biol Res Nurs. 2010 Jul;12(1):28-36. doi: 10.1177/1099800410361535. Epub 2010 May 7. PMID 20453024
- [Background] Epstein M, Preston S, Weitzman RE. Isoosmotic central blood volume expansion suppresses plasma arginine vasopressin in normal man. J Clin Endocrinol Metab. 1981 Feb;52(2):256-62. doi: 10.1210/jcem-52-2-256. PMID 7007402
- [Background] Farhi LE, Linnarsson D. Cardiopulmonary readjustments during graded immersion in water at 35 degrees C. Respir Physiol. 1977 Jun;30(1-2):35-50. doi: 10.1016/0034-5687(77)90020-2. PMID 877449
- [Background] Hammerum MS, Bie P, Pump B, Johansen LB, Christensen NJ, Norsk P. Vasopressin, angiotensin II and renal responses during water immersion in hydrated humans. J Physiol. 1998 Aug 15;511 ( Pt 1)(Pt 1):323-30. doi: 10.1111/j.1469-7793.1998.323bi.x. PMID 9679185
- [Background] Johansen LB, Jensen TU, Pump B, Norsk P. Contribution of abdomen and legs to central blood volume expansion in humans during immersion. J Appl Physiol (1985). 1997 Sep;83(3):695-9. doi: 10.1152/jappl.1997.83.3.695. PMID 9292451
- [Background] Nater UM, La Marca R, Florin L, Moses A, Langhans W, Koller MM, Ehlert U. Stress-induced changes in human salivary alpha-amylase activity -- associations with adrenergic activity. Psychoneuroendocrinology. 2006 Jan;31(1):49-58. doi: 10.1016/j.psyneuen.2005.05.010. Epub 2005 Jul 5. PMID 16002223
- [Background] Nater UM, Rohleder N, Schlotz W, Ehlert U, Kirschbaum C. Determinants of the diurnal course of salivary alpha-amylase. Psychoneuroendocrinology. 2007 May;32(4):392-401. doi: 10.1016/j.psyneuen.2007.02.007. Epub 2007 Apr 5. PMID 17418498
- [Background] Petrakova L, Doering BK, Vits S, Engler H, Rief W, Schedlowski M, Grigoleit JS. Psychosocial Stress Increases Salivary Alpha-Amylase Activity Independently from Plasma Noradrenaline Levels. PLoS One. 2015 Aug 6;10(8):e0134561. doi: 10.1371/journal.pone.0134561. eCollection 2015. PMID 26247781
- [Background] de Kloet CS, Vermetten E, Geuze E, Wiegant VM, Westenberg HG. Elevated plasma arginine vasopressin levels in veterans with posttraumatic stress disorder. J Psychiatr Res. 2008 Feb;42(3):192-8. doi: 10.1016/j.jpsychires.2006.11.009. Epub 2007 Jan 11. PMID 17222428